CLINICAL TRIAL: NCT01956344
Title: Neural Mechanisms of CBT Response in Hoarding Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Tolin, Dr, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01MH101163-01 (NIH); 1R01MH101163-01 (NIH)
Record Dates: First submitted 2013-09-12; First posted 2013-10-08 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Hoarding Disorder; Clutter; CBT; Cognitive behavior therapy; fMRI; Obsessive compulsive disorder (OCD); Healthy control
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Hoarding Disorder; Speech Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Immediate Treatment (Experimental): Cognitive-behavioral therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Delayed Treatment (No Intervention): This group will receive the cognitive-behavioral therapy after a 16 week delay
- Healthy Control (No Intervention): This group is matched to the immediate treatment group on age and gender. They do not receive an active treatment and will be used a a healthy comparator group.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Group cognitive-behavioral therapy for hoarding disorder, 16 weeks
  Arms: Immediate Treatment

SUMMARY:
The purpose of this research is to measure changes in brain activity with functional magnetic resonance imaging (fMRI) before and after cognitive-behavioral therapy for compulsive hoarding. Cognitive-behavioral therapy aims to help people change the thoughts and behaviors that maintain symptoms of hoarding. The investigators intend to enroll approximately 80 people with hoarding disorder and 40 people with no psychiatric disorder, between the ages of 20 and 60, for this study. The investigators believe that after treatment there will be changes in the brain activity of individuals with compulsive hoarding.

DETAILED DESCRIPTION:
The long-term goal of the proposed research is to improve clinical outcomes for Hoarding Disorder (HD), a common and potentially debilitating condition that poses a severe public health burden. The PI has developed and tested a cognitive-behavioral therapy (CBT) that appears moderately effective, although there is clear room for improvement. In the present study, the investigators propose to merge this line of research with the PI's recent NIH-supported neuroimaging research that points to specific functional abnormalities in regions of interest (ROIs) related to cognitive and affective decisionmaking processes. Patients with HD n = 80) will be randomized to CBT or wait list (WL). At pre-treatment, mid-treatment, and post-treatment, patients will undergo functional magnetic resonance imaging (fMRI) during an acquiring and discarding decision-making task that has been used successfully in the investigators' previous work. In addition, patients will complete a number of laboratory tasks designed to assess decision-making capacity and impairment. A group of healthy control (HC) participants (n = 40) will also complete these measures as a normative control group. The primary aim of the proposed study is to determine the extent to which the observed patterns of neural activity in HD change following CBT. Under this aim, the investigators predict that HD patients (vs.HCs) will show greater hemodynamic activity in ROIs associated with cognitive and affective aspects of decision-making. The investigators further predict that HD patients receiving CBT (vs. WL) will show decreased activity in those ROIs, and will no longer differ from HCs following CBT. A secondary aim of the proposed study is to determine the relationship between change in activity in brain regions of interest and hoarding-related symptoms and impairments. The investigators expect, that hemodynamic activity in the target ROIs will correlate with symptoms of HD and with performance on decision-making tasks; and that change in brain activity will correspond to both symptom and mechanism changes over the course of treatment. Finally, an exploratory aim is to explore, using both data-driven and model-constrained approaches, patterns of pre-treatment neural activity that predict response to CBT. The investigators predict that among treated HD patients, pre-treatment activity in the target ROIs will correlate significantly with HD symptom change from pre- to posttreatment. Results of the proposed study are expected to elucidate the neural mechanisms of successful response to CBT treatment for hoarding patients, and to set the stage for further treatment development and possible improvements in outcome for this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-65
* Hoarding Disorder primary condition
* Score at least 4 on the CGI
* Free from all psychotropic medications for at least 4 weeks(5 weeks for fluoxetine)
* Participant is fluent in English
* Control over current living environment (i.e. not living in a nursing home or with relatives)
* Physically able to complete therapy assignments (i.e able to discard etc)
* Able to complete study measures
* If female: Using an approved method of contraception

Exclusion Criteria:

* More than 10 sessions of CBT for HD
* Actively suicidality, previous suicide attempt, current use of self harming behaviors or is at risk for harming others
* Current or past diagnosis of serious psychological disorder (psychotic disorder, bipolar disorder, substance use disorder or uncontrolled anorexia)
* Psychiatric hospitalization within the past 12 months
* History of anoxic or traumatic brain injury
* Evidence of cognitive dysfunction that would interfere in the ability to provide informed consent or engage in CBT
* Claustrophobia
* Pacemaker, aneurysm clip, or other metal in the body that would pose a risk during fMRI?
* If female: Pregnant or lactating

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Saving Inventory-Revised (SI-R) | Change from baseline at 8 weeks and 16 weeks after treatment
  The SI-R is a 23-item questionnaire with 3 factor-analytically defined sub-scales for difficulty discarding, excessive clutter and compulsive acquisition

SECONDARY OUTCOMES:
Clinician Global Impression (CGI) Severity (Self Report and Clinician Administered) | Change from baseline at 8 weeks and 16 weeks after treatment
  The CGI is a widely used measure of global symptom severity (CGI-S) and symptom improvement after treatment (CGI-I). On the CGI-S the scale ranges from 1 (no symptoms) to 7 (extreme symptoms). On the CGI-I the scale ranges from 1 (very much improved) to 7 (very much worse). The CGI can be used in both a self-report and clinician administered version and this study utilizes both formats.

CONTACTS AND LOCATIONS:
Overall Officials: David F Tolin, Ph.D., Principal Investigator — Anxiety Disorders Center, Institute of Living
Locations (1):
- Anxiety Disorders Center, Institute of Living, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
We will upload de-identified study data to an online database to be shared with colleagues upon request.

REFERENCES:
- [Derived] Tolin DF, Levy HC, Hallion LS, Wootton BM, Jaccard J, Diefenbach GJ, Stevens MC. Changes in neural activity following a randomized trial of cognitive behavioral therapy for hoarding disorder. J Consult Clin Psychol. 2023 Apr;91(4):242-250. doi: 10.1037/ccp0000804. Epub 2023 Mar 6. PMID 36877480
- [Derived] Wootton BM, Bragdon LB, Worden BL, Diefenbach GJ, Stevens MC, Tolin DF. Measuring Within-Session and Between-Session Compliance in Hoarding Disorder: A Preliminary Investigation of the Psychometric Properties of the CBT Compliance Measure (CCM) and Patient Exposure/Response Prevention Adherence Scale for Hoarding (PEAS-H). Assessment. 2021 Sep;28(6):1694-1707. doi: 10.1177/1073191120918024. Epub 2020 May 2. PMID 32362128
- [Derived] Stevens MC, Levy HC, Hallion LS, Wootton BM, Tolin DF. Functional Neuroimaging Test of an Emerging Neurobiological Model of Hoarding Disorder. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Jan;5(1):68-75. doi: 10.1016/j.bpsc.2019.08.010. Epub 2019 Sep 5. PMID 31676206
- [Derived] Tolin DF, Wootton BM, Levy HC, Hallion LS, Worden BL, Diefenbach GJ, Jaccard J, Stevens MC. Efficacy and mediators of a group cognitive-behavioral therapy for hoarding disorder: A randomized trial. J Consult Clin Psychol. 2019 Jul;87(7):590-602. doi: 10.1037/ccp0000405. Epub 2019 Apr 22. PMID 31008633
- [Derived] Levy HC, Katz BW, Das A, Stevens MC, Tolin DF. An investigation of delay and probability discounting in hoarding disorder. J Psychiatr Res. 2019 Feb;109:89-95. doi: 10.1016/j.jpsychires.2018.11.019. Epub 2018 Nov 22. PMID 30513489
- [Derived] Tolin DF, Hallion LS, Wootton BM, Levy HC, Billingsley AL, Das A, Katz BW, Stevens MC. Subjective cognitive function in hoarding disorder. Psychiatry Res. 2018 Jul;265:215-220. doi: 10.1016/j.psychres.2018.05.003. Epub 2018 May 4. PMID 29751168